CLINICAL TRIAL: NCT04189705
Title: A Multi-center, Randomized, Double-blind, Active-controlled, Non-inferiority, Phase 3 Study to Evaluate the Efficacy and Safety of MCT-SR in Patients With Gastritis
Brief Title: A Study to Evaluate the Efficacy and Safety of MCT-SR in Patients With Gastritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 037-402-00039
Record Dates: First submitted 2019-11-25; First posted 2019-12-06 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Acute Gastritis; Chronic Gastritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MCT-SR (Experimental): Drug: MCT-SR 2 times/day for 2 weeks
  Interventions: Drug: MCT-SR; Drug: Mucosta Tab.
- Mucosta Tab. (Active Comparator): Drug: Mucosta Tab. 3 times/day for 2 weeks
  Interventions: Drug: MCT-SR; Drug: Mucosta Tab.

INTERVENTIONS:
Drug: MCT-SR — Rebamipide 150mg
Drug: Mucosta Tab. — Rebamipide 100mg
  Other Names: Mucosta

SUMMARY:
This is a multi-center, randomized, double-blind, active-controlled, non-inferiority, phase 3 study to evaluate the efficacy and safety of MCT-SR in patients with gastritis.

DETAILED DESCRIPTION:
To contribute greater treatment compliance and patient convenience, the rebamipide SR formulation has been developed.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females aged ≥19 and <75 years
* Patients diagnosed with acute or chronic gastritis by gastroscopy with at least 1 erosion confirmed by gastroscopy within 7 days prior to the first dose of the Investigational Product(IP)

Exclusion Criteria:

* Patients ineligible for gastroscopy
* Patients who took other drugs for treating gastritis within 2 weeks prior to the first dose of the IP.
* Patients who have to continue taking drugs that may induce gastritis
* Other clinically significant medical or psychiatric findings that the investigator considers inappropriate for the study

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2020-04-23 (Actual); Study Completion 2020-04-23 (Actual)

PRIMARY OUTCOMES:
Endoscopic Improvement Rate | 2 weeks
  The percentage of subjects with improvement refer to those with more than 50% improvement in erosion score on gastroscopy after treatment compared to the score before treatment.

CONTACTS AND LOCATIONS:
Overall Officials: JaeGyu Kim, Ph.D., Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Locations (1):
- Chung-Ang University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No